CLINICAL TRIAL: NCT03446807
Title: Safety and Efficacy of Droxidopa for Fatigue in Patients With Parkinsonism
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision to terminate
Sponsor: Loma Linda University (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5170406
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Parkinson Disease; Multiple System Atrophy; Progressive Supranuclear Palsy
Keywords: fatigue; Droxidopa
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive; Fatigue | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The first phase is double-blind and the second phase is open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Droxidopa (Experimental): The Droxidopa starting dose for all eligible patients in the Titration Periods are 100mg three times daily (TID). Doses will be titrated by 100mg TID; increments will be made weekly until the optimal dose is achieved or the subject doesn't notice an improvement in their subjective fatigue on a higher dose compared to the most recent dose. Half of the subjects will be on Droxidopa for 3 months during the double-blind phase. All subjects will be on Droxidopa for 3 months during the open-label phase.
  Interventions: Drug: Droxidopa
- Placebo Oral Tablet (Placebo Comparator): The placebo starting dose for all eligible patients in the Titration Period is 100mg TID. Doses will be titrated by 100mg TID; increments will be made weekly until the optimal dose is achieved. Half of the subjects will be on placebo for 3 months during the double-blind phase.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Droxidopa — Droxidopa in 100, 200, and 300mg capsules. Maximum dose to be used in this study is 600mg.
  Other Names: Northera
  Arms: Droxidopa
Drug: Placebo Oral Tablet — Placebo capsules to match Droxidopa 100, 200, and 300mg capsules.
  Other Names: Placebo
  Arms: Placebo Oral Tablet

SUMMARY:
The purpose of this study is to determine the efficacy of Droxidopa for the treatment of fatigue in patients with Parkinsonism by the Visual Analog Fatigue Scale (VAFS). This is a randomized, placebo-controlled, double-blind clinical trial for 3 months where half the subjects will receive placebo and the other half will receive Droxidopa. Following this will be a wash-out period of 7 days and then all subjects will receive Droxidopa for 3 months during the open-label phase.

DETAILED DESCRIPTION:
Parkinsonism, is a group of symptoms seen in several diseases, including Parkinson's Disease. In Parkinsonism, a patient may become stiff, have smaller and slower movements, develop a tremor (shaking of the arms or legs), have decreased facial expression, and a softer voice.

Fatigue is a common symptom that causes suffering and stress in diseases that affect the brain. Over 50% of patients with Parkinsonism report fatigue as one of their top three symptoms that make their life more difficult. Currently, there are no evidence-based guidelines for treating fatigue in Parkinson's Disease, and no effective medications or therapeutic modalities exist for fatigue symptoms in patients with Parkinson's Disease.

Droxidopa (also known by the trade name NORTHERA) is a safe and well tolerated medication which has been approved in USA for the treatment of orthostatic dizziness or light headedness in patients with a clinical diagnosis of symptomatic Neurogenic Orthostatic Hypotension associated with primary autonomic failure (Parkinson's Disease and Multiple System Atrophy), Dopamine Beta Hydroxylase Deficiency, or Non Diabetic Autonomic Neuropathy.

Fatigue may be due to diminished levels of norepinephrine in Parkinson's Disease. The locus coeruleus, one of the major sources of norepinephrine, is affected during the preclinical phase of Parkinson's Disease during stage 2 of Braak pathology staging. Norepinephrine is the final metabolite of dopamine, therefore by adding exogenous norepinephrine, it may be possible to control some of the motor and non-motor symptoms of Parkinsonism. Norepinephrine is the final metabolite of droxidopa, and it is still unclear if it passes the blood-brain barrier. This pilot study is to measure the efficacy and safety of droxidopa in Parkinsonism patients with fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Age of 50 years or older.
* Clinical diagnosis of Parkinsons Disease or Atypical Parkinsonism (including multiple system atrophy (MSA), PSP)
* Fluent in English
* Reported fatigue and must have a mean VAFS score of 4 or more at baseline
* Written informed consent

Exclusion Criteria:

* Inability to understand or cooperate with study procedures
* Alcohol or substance use disorder within the past 12 months (as per Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria)
* Women who are pregnant or breastfeeding
* Women of childbearing potential (WOCP) as indicated by one of the following:
* Sustained supine hypertension greater than or equal to 180 mmHg systolic or 110 mmHg diastolic. Sustained is defined as the average of 3 observations each at least 10 minutes apart with the patient having been supine and at rest for at least 5 minutes prior to each measurement
* Untreated closed angle glaucoma
* Diagnosis of hypertension that requires treatment with antihypertensive medications
* Any significant uncontrolled cardiac arrhythmia
* History of myocardial infarction, within the past 2 years
* Current unstable angina
* Congestive heart failure (NYHA Class 3 or 4)
* Diabetic autonomic neuropathy
* History of cancer within the past 2 years other than a successfully treated, non-metastatic cutaneous squamous cell or basal cell carcinoma or cervical cancer in situ
* Gastrointestinal condition that may affect the absorption of Investigational Medicinal Product (e.g. ulcerative colitis, gastric bypass)
* Any major surgical procedure within 30 days prior to the first titration visit.
* Currently receiving any investigational drug or have received an investigational drug within 28 days prior to the first titration visit
* Any condition or laboratory test result, which in the Investigator's judgment, might result in an increased risk to the patient, or would affect their participation in the study
* Dementia or non-treated depression
* Subjects who have a mean VAFS score of less than 4 at baseline
* Vulnerable populations
* Uncontrolled intercurrent illnesses including, but not limited to severe lung disease, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia, and situations that would limit compliance with study requirements will be excluded
* Orthostatic hypotension (OH)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Droxidopa on fatigue in subjects with Parkinsonism as determined by completion of Visual Analogue Fatigue Scale (VAFS) | Change between baseline and 12 weeks
  Subjects will complete the VAFS which measures level of fatigue with zero being equivalent to energetic with no fatigue to ten being worst possible fatigue
Efficacy of Droxidopa on fatigue in subjects with Parkinsonism as determined by completion of Visual Analogue Fatigue Scale (VAFS) | Change between 18 weeks and 28 weeks
  Subjects will complete the VAFS which measures level of fatigue with zero being equivalent to energetic with no fatigue to ten being worst possible fatigue
Efficacy of Droxidopa on fatigue in subjects with Parkinsonism as determined by completion of Visual Analogue Fatigue Scale (VAFS) | Week 29
  Subjects will complete the VAFS which measures level of fatigue with zero being equivalent to energetic with no fatigue to ten being worst possible fatigue

SECONDARY OUTCOMES:
Efficacy of Droxidopa on motor and non-motor symptoms of Parkinsonism as determined by the Unified Parkinson's Disease Rating Scale (UPDRS) | Change between baseline and 12 weeks
  The UPDRS is a composite measurement of motor and non-motor symptoms divided into six domains. Domain I measures Mentation, Behavior and Mood. Domain II measures Activities of Daily Living. Domain III measures Motor Examination. Domain IV measures Complications of Therapy. Domain V is Modified Hoehn and Yahr Staging. Domain 6 is Schwab and England Activities of Daily Living Scale
Efficacy of Droxidopa on motor and non-motor symptoms of Parkinsonism as determined by the Unified Parkinson's Disease Rating Scale (UPDRS) | Change between 18 weeks and 28 weeks
  The UPDRS is a composite measurement of motor and non-motor symptoms divided into six domains. Domain I measures Mentation, Behavior and Mood. Domain II measures Activities of Daily Living. Domain III measures Motor Examination. Domain IV measures Complications of Therapy. Domain V is Modified Hoehn and Yahr Staging. Domain 6 is Schwab and England Activities of Daily Living Scale
Efficacy of Droxidopa on motor and non-motor symptoms of Parkinsonism as determined by the Unified Parkinson's Disease Rating Scale (UPDRS) | Week 29
  The UPDRS is a composite measurement of motor and non-motor symptoms divided into six domains. Domain I measures Mentation, Behavior and Mood. Domain II measures Activities of Daily Living. Domain III measures Motor Examination. Domain IV measures Complications of Therapy. Domain V is Modified Hoehn and Yahr Staging. Domain 6 is Schwab and England Activities of Daily Living Scale

CONTACTS AND LOCATIONS:
Overall Officials: Khashayar Dashtipour, M.D. Ph.D., Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Faculty Medical Offices - Neurology Clinic, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Lundbeck is funding this study and will be providing the study drug. If Lundbeck requests, they will be provided with protocol, statistical analysis plan, clinical study report, and any other study data they request. All adverse events will be reported to Lundbeck.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available to Lundbeck from the start of the study through it's completion.
Access Criteria: This material will be provided to Lundbeck in person, not electronically.

REFERENCES:
- [Background] Friedman J, Friedman H. Fatigue in Parkinson's disease. Neurology. 1993 Oct;43(10):2016-8. doi: 10.1212/wnl.43.10.2016. PMID 8413960
- [Background] Friedman JH, Brown RG, Comella C, Garber CE, Krupp LB, Lou JS, Marsh L, Nail L, Shulman L, Taylor CB; Working Group on Fatigue in Parkinson's Disease. Fatigue in Parkinson's disease: a review. Mov Disord. 2007 Feb 15;22(3):297-308. doi: 10.1002/mds.21240. PMID 17133511
- [Background] Friedman JH, Beck JC, Chou KL, Clark G, Fagundes CP, Goetz CG, Herlofson K, Kluger B, Krupp LB, Lang AE, Lou JS, Marsh L, Newbould A, Weintraub D. Fatigue in Parkinson's disease: report from a mutidisciplinary symposium. NPJ Parkinsons Dis. 2016;2:15025-. doi: 10.1038/npjparkd.2015.25. Epub 2016 Jan 14. PMID 27239558
- [Background] Mendonca DA, Menezes K, Jog MS. Methylphenidate improves fatigue scores in Parkinson disease: a randomized controlled trial. Mov Disord. 2007 Oct 31;22(14):2070-6. doi: 10.1002/mds.21656. PMID 17674415
- [Background] Smith KM, Eyal E, Weintraub D; ADAGIO Investigators. Combined rasagiline and antidepressant use in Parkinson disease in the ADAGIO study: effects on nonmotor symptoms and tolerability. JAMA Neurol. 2015 Jan;72(1):88-95. doi: 10.1001/jamaneurol.2014.2472. PMID 25420207
- [Background] Kaufmann H, Freeman R, Biaggioni I, Low P, Pedder S, Hewitt LA, Mauney J, Feirtag M, Mathias CJ; NOH301 Investigators. Droxidopa for neurogenic orthostatic hypotension: a randomized, placebo-controlled, phase 3 trial. Neurology. 2014 Jul 22;83(4):328-35. doi: 10.1212/WNL.0000000000000615. Epub 2014 Jun 18. PMID 24944260
- [Background] Herlofson K, Larsen JP. Measuring fatigue in patients with Parkinson's disease - the Fatigue Severity Scale. Eur J Neurol. 2002 Nov;9(6):595-600. doi: 10.1046/j.1468-1331.2002.00444.x. PMID 12453074
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775

DOCUMENTS (1):
  • Study Protocol (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03446807/Prot_000.pdf